CLINICAL TRIAL: NCT06542432
Title: A Prospective Trial to Assess Clinical Utility and Effectiveness of MyOme's Polygenic Risk Score for Coronary Artery Disease (COMPASS-CAD)
Brief Title: Utility and Effectiveness of Polygenic Risk Scoring (PRS) for Coronary Artery Disease (CAD)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: MyOme (Industry)
Collaborators: University of Pennsylvania (Other); Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 004
Record Dates: First submitted 2024-03-29; First posted 2024-08-07 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease; Polygenic Risk Score; Heart Diseases; Coronary Disease; Myocardial Infarction; Cardiovascular Diseases
Keywords: Polygenic risk score; Integrated risk score; Genetics; Cardiovascular health; Coronary artery disease; Precision medicine
MeSH Terms: conditions — Coronary Artery Disease; Genetic Risk Score; Heart Diseases; Coronary Disease; Myocardial Infarction; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Intervention (Experimental): Participants will receive their integrated risk score result for coronary artery disease.
  Interventions: Genetic: Disclosure of integrate risk score for coronary artery disease
- No Intervention: Control (No Intervention): Participants will only receive standard of care ASCVD Pooled Cohorts Equation (ASCVD PCE), and disclosure of integrated risk score result will be deferred until 3 years after enrollment.

INTERVENTIONS:
Genetic: Disclosure of integrate risk score for coronary artery disease — Participants will receive their integrated risk score for coronary disease along with an optional genetic counseling visit to discuss the results.
  Arms: Experimental: Intervention

SUMMARY:
The goal of this study is to assess the benefit to physicians and patients of adding an integrated risk score (IRS) to existing coronary artery risk tools by conducting a randomized prospective study. IRS combines both an individual's coronary artery disease (CAD) polygenic risk score (PRS) and clinical risk factors, like cholesterol levels and age. This study will examine to what extent IRS knowledge impacts physician/provider behavior as well as clinical outcomes including cholesterol levels and incident heart disease.

DETAILED DESCRIPTION:
This is a 1:1 randomized controlled trial of participants with no known coronary artery disease, are not on lipid-lowering therapy, and do not have LDL-C over 190mg/dL. Participants will be recruited from cohorts that have been previously genotyped and found to have either elevated or average risk based on a CAD IRS. Participants will be randomized into two equal groups: one group will receive their IRS result for coronary artery disease at baseline, and the other group will receive their ASCVD Pooled Cohorts Equation result at baseline and CAD IRS result approximately 3 years after enrollment. Subject data will be collected for 5 years from the time of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* ASCVD risk ≥5% and below 20% over the following 10 years as defined by the standard pooled cohort equations
* No previous CAD event (inclusive of myocardial infarction, diagnosis of CAD, stroke)
* Previously genotyped as part of a research study that enables recontact of participants
* Receiving primary care at a participating institution.

Exclusion Criteria:

* Prior diagnosis of CAD: inclusive of prior myocardial infarction and revascularization (stent or coronary artery bypass grafting)
* Currently treated with lipid-lowering therapy, including statins, ezetimibe, PCSK9 inhibitors, inclisiran, or bempedoic acid
* Future use of statins contraindicated
* Prior diagnosis of Cerebrovascular disease: Inclusive of history of ischemic stroke, transient ischaemic attack (TIA), carotid endarterectomy, carotid artery stenting
* Prior diagnosis of Peripheral arterial disease: Inclusive of history of claudication, revascularization (stents or bypass)
* Severe hypercholesterolemia (LDL-C ≥ 190 mg/dL)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Does receiving an IRS report influence clinical decision making, including the provider's decision to treat with lipid lowering medication or order diagnostic testing? | 5 years
  Aggregating longitudinal clinical data will be collected to compare the incidence of lipid-lowering medication initiation and cardiac diagnostic testing between the intervention arm which received their integrated risk score and the control group.
Does receiving an IRS report affect patient clinical measurements, including LDL-C levels? | 5 years
  Aggregating longitudinal clinical data will be collected to compare the clinical measurements between the intervention arm which received their integrated risk score and the control group.

SECONDARY OUTCOMES:
Does the IRS identify those at elevated risk for CAD and future ASCVD events? | 5 years
  Aggregated longitudinal clinical data and patient survey data will be collected to compare patient clinical outcomes in those with a high CAD IRS.
Does receiving an IRS report affect the incidence of CAD events? | 5 years
  Aggregated longitudinal clinical data will be collected to compare patient clinical outcomes in those with a CAD IRS reported at baseline and the control group.
Does receiving an IRS report affect participant understanding of their individual CAD risk? | 5 years
  Patient survey data will be collected to assess their understanding of their CAD risk.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - University of Pennsylvania, Philadelphia, Pennsylvania